CLINICAL TRIAL: NCT02614313
Title: Assessment of Psychological and Metabolic Responses During Fructose Intolerance Breath Tests in Patients With Functional GI Disorders: Placebo-controlled Breath Testing
Brief Title: Fructose Breath-testing in Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brain-Gut Research Group (Other)
Collaborators: New Jersey Medical School (Other); National University of Singapore (Other)
Responsible Party: Principal Investigator, C. Wilder-Smith, Dr., Brain-Gut Research Group
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: BGRG FBT-PLA
Record Dates: First submitted 2015-11-16; First posted 2015-11-25 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Functional Gastrointestinal Disorders; Irritable Bowel Syndrome
Keywords: Fructose; Irritable Bowel Syndrome; Breath test; Placebo
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome | interventions — Fructose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fructose double-blind (Active Comparator): Fructose during breath test, double-blind 35g
  Interventions: Procedure: Blinded breath test with fructose
- Fructose open (Active Comparator): Fructose during breath test, open 35g
  Interventions: Procedure: Open breath test with fructose
- Sweet placebo double-blind (Placebo Comparator): Assugrin during breath test double-blind
  Interventions: Procedure: Breath test with sweet placebo (Assugrin)
- Neutral placebo double-blind (Placebo Comparator): Water during breath test double-blind
  Interventions: Procedure: Breath test with neutral placebo (still water)

INTERVENTIONS:
Procedure: Open breath test with fructose — Open randomised fructose 35g during breath test
  Arms: Fructose open
Procedure: Breath test with sweet placebo (Assugrin) — Double-blind randomised breath-testing with sweet placebo (Assugrin)
  Arms: Sweet placebo double-blind
Procedure: Breath test with neutral placebo (still water) — Double-blind randomised breath-testing with neutral placebo
  Arms: Neutral placebo double-blind
Procedure: Blinded breath test with fructose — Double-blind randomised fructose 35g during breath test
  Arms: Fructose double-blind

SUMMARY:
Background: Breath testing for food intolerances is becoming routine in patients with functional gastrointestinal disorders (FGID). Both FGID and saccharide intolerances (FODMAPs: fermentable oligo-, di-, polysaccharide and polyols, e.g. lactose, fructose, sorbitol) are common (>10% of any given population) and often respond to dietary modification. The breath tests are based on quantification of gas excretion in breath as a sign of malabsorption and symptom provocation, but are likely subject to considerable psychological bias. The role of expectation and other psychological effects on breath testing has not been reported, but is crucial for the validation of these increasingly wide-spread tests with considerable dietary and potentially deleterious consequences. Fructose has been shown to result in short term pro-inflammatory metabolic responses, but these effects have not been studied as underlying causes for intolerance symptoms in fructose intolerant patients with FGID.

Aim: To investigate the psychological component and the short-term metabolic effects of fructose breath testing in patients referred for evaluation of FGID using placebo. Additionally, to assess baseline predictors for a positive breath test result.

Methods: Fructose intolerance (defined by a positive symptom index) and malabsorption (defined by increased breath hydrogen/methane concentrations) will be determined in 30 successive male and female FGID in a single centre using breath-testing. Fructose 35g, given double-blind as well as open, a sweet placebo (cyclamate/saccharine; Assugrin®) and a neutral (still water) placebo given double-blind will be compared in a randomized, cross-over sequence and according to our standardised procedure on four separate study days. Symptoms will be recorded using standardised questionnaires and breath concentrations of H2 and CH4 will be measured during testing on the four study days. Somatisation and psychological profiles will be assessed by questionnaires. Blood samples will be obtained before and during provocation testing to assess short-term responses to fructose loading by metabolomics. Fructose, blinded and open, and placebo responses will be compared and baseline predictors for a positive breath tests assessed.

ELIGIBILITY:
Inclusion criteria

* Thirty male or female FGID (Irritable Bowel Syndrome or Functional Dyspepsia according to the Rome III criteria) patients -
* 10 healthy female and male controls
* aged between 18 and 60 years

Exclusion criteria:

* Bowel resections, except appendicectomy or cholecystectomy
* Evidence of organic disease
* No medications (excluding antihypertensives, antidepressants and low-dose aspirin), including herbal, from 4 days before the first study day until after breath test
* Coeliac's disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Fructose intolerance, as percentage of patients | 5 hours
  Defined by symptom scores

SECONDARY OUTCOMES:
Between-group comparisons of breath test gas concentrations and symptom indices | 5 hours
  Breath gas concentrations and cumulative symptoms experienced during breath testing will be compared between treatment groups
Correlations between breath test gas concentrations, symptom indices and metabolite | 5 hours
  Correlations between changes in gas levels, GI symptoms from baseline and changes in metabolites identified by metabolomic analysis in the different treatment and responder groups (i.e intolerance or no intolerance as defined by the standard breath test results). Metabotype and psychological predictors at baseline for intolerance (responder) status during breath testing will be assessed by multiple regression analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastoenterology Group Practice, Bern, Switzerland